CLINICAL TRIAL: NCT01865110
Title: Efficacy of Alternating Immunochemotherapy Consisting of R-CHOP + R-HAD vs R-CHOP Alone, Followed by Maintenance Therapy Consisting of Additional Lenalidomide + Rituximab vs Rituximab Alone for Older Patients With Mantle Cell Lymphoma
Brief Title: R-CHOP + R-HAD vs R-CHOP Followed by Maintenance Lenalidomide + Rituximab vs Rituximab for Older Patients With MCL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCL R2 Elderly
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; RCHOP; RHAD; rituximab; lenalidomide
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — R-CHOP protocol; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Induction experimental arm (Experimental): R-CHOP / R-HAD : Alternating 3 cycles of R-CHOP administered in 3 week cycles + 3 cycles of R-HAD administered in 4 week cycles.
  Interventions: Drug: R-CHOP / R-HAD
- Standart induction arm (Active Comparator): 8 cycles of R-CHOP administered in 3 week cycles
  Interventions: Drug: R-CHOP
- Maintenance experimental arm (Experimental): lenalidomide + rituximab : 13 cycles of rituximab SC 1400 mg administered in 8 week cycles + 26 cycles Lenalidomide 15 mg 3 weeks every 4 weeks for 24 months
  Interventions: Drug: Rituximab; Drug: Lenalidomide
- Maintenance standart arm (Active Comparator): 13 cycles of rituximab SC 1400 mg administered in 8 week cycles for 24 months
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: R-CHOP — R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone) administered in 3 week cycles for 8 cycles
  Other Names: rituximab, CHOP
  Arms: Standart induction arm
Drug: R-CHOP / R-HAD — R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) administered in 3 week cycles for 3 cycles R-HAD (rituximab, cytarabine, dexamethasone) administered in 3 week cycles for 4 cycles alternating
  Other Names: rituximab, CHOP; rituximab HD AraC
  Arms: Induction experimental arm
Drug: Rituximab — Rituximab SC 1400 mg every 8 weeks for 24 months
  Other Names: Mabthera
  Arms: Maintenance experimental arm; Maintenance standart arm
Drug: Lenalidomide — Lenalidomide 15 mg 3 weeks every 4 weeks for 24 months
  Other Names: Revlimid
  Arms: Maintenance experimental arm

SUMMARY:
This study aims to evaluate whether the addition of lenalidomide to rituximab-maintenance improves progression free survival (PFS) compared to standard rituximab maintenance after induction treatment consisting of R-CHOP + R-HAD vs R-CHOP alone in older patients (≥ 60 year old) with mantle cell lymphoma.

The treatments consist of two phases: induction treatment (3 R-CHOP21 + 3 cycles of R-HAD28 alternating) vs 8 cycles of R-CHOP21) followed by maintenance treatment (13 cycles of rituximab + 26 cycles of lenalidomide vs 13 cycles of rituximab).

DETAILED DESCRIPTION:
This study aims to evaluate whether the addition of lenalidomide to rituximab-maintenance improves progression free survival (PFS) compared to standard rituximab maintenance after induction treatment consisting of R-CHOP + R-HAD versus R-CHOP alone in older patients (≥ 60 year old) with mantle cell lymphoma. 643 patients will be randomized in induction phase and 433 in maintenance phase.

The treatments consist of two phases:

* induction treatment will be 3 cycles of R-CHOP21 + 3 cycles of R-HAD28(alternating) versus 8 cycles of R-CHOP21 alone
* maintenance treatment will be 13 cycles of rituximab every 8 weeks + 26 cycles of lenalidomide every 4 weeks vs 13 cycles of rituximab every 8 weeks.

Patients will be followed 2.5 years after the last patient randomized for maintenance for final analysis. All subjects who complete or discontinue the maintenance treatment for any reason will be followed for at least 3 years after his/her last study treatment administration in maintenance period for Second Primary Malignancies (SPM). A long term follow-up for progression/death will be done up to the end of period of SPM data collection.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent form Biopsy-proven MCL according to WHO classification

≥ 60 years of age and ineligible for autologous transplant Ann Arbor stage II-IV Previously untreated ECOG PS ≤ 2

Male subjects must:

* agree to use a condom during sexual contact with a woman of childbearing potential, even if they have had a vasectomy, throughout lenalidomide therapy
* agree to not donate semen during lenalidomide therapy.

All subjects must:

* have an understanding that the lenalidomide could have a potential teratogenic risk.
* agree to abstain from donating blood while taking lenalidomide therapy
* agree not to share study medication with another person.
* be counselled about pregnancy precautions and risks of foetal exposure.

Additional criteria for randomization in maintenance phase:

* CR, CRu or PR after induction treatment, determined as per Cheson 1999 criteria
* During the run-in period of 6 months starting from the date of the first randomization in the trial: in case of direct randomization into maintenance phase, patient must have been treated in first line by 6-8 cycles of R-CHOP.

Exclusion Criteria:

Female of childbearing potential

Any of the following laboratory abnormalities at diagnosis, if not related to lymphoma:

Absolute neutrophils count <1,000 /mm3 Platelet count < 75,000/mm3 AST/SGOT or ALT/SGPT >3.0 UNL Serum total bilirubin > 1.5 ULN (except if due to Gilbert's syndrome) Calculated creatinine clearance (Cockcroft-Gault formula or MDRD) < 30 mL / min Central Nervous System involvement by lymphoma Contraindication for medical DVT prophylaxis for patients at high risk for DVT

Prior history of malignancies other than MCL unless the subject has been free of the disease for ≥ 5 years. Exceptions include the following:

* Basal cell carcinoma or Squamous cell carcinoma of the skin
* Carcinoma in situ of the cervix or of the breast
* Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b). Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent the patient to receive the study medication as planned.

Seropositivity for human immunodeficiency virus at study entry Seropositivity for hepatitis C virus at study entry,

Active viral infection with hepatitis B virus at study entry:

* HBsAg positive
* HBsAg negative, anti-HBs positive and anti-HBc positive

Uncontrolled illness including, but not limited to:

* Active infection requiring parenteral antibiotics.
* Uncontrolled diabetes mellitus
* Chronic symptomatic congestive heart failure (Class NYHA III or IV).
* Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
* Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia.

Prior ≥ Grade 3 allergic hypersensitivity to thalidomide. Prior ≥ Grade 3 rash or any desquamating (blistering) rash while taking thalidomide.

Known anti-murine antibody (HAMA) reactivity or known hypersensitivity to murine antibodies.

Subjects with ≥ Grade 2 neuropathy. Prior use of lenalidomide Participation in another clinical trial within three weeks before randomization in this study

Additional criteria for randomization in maintenance phase:

* SD or PD after induction treatment determined as per Cheson 1999 criteria
* Patient treated by induction immuno-chemotherapy other than 6-8 cycle of R-CHOP21 or 2-3 cycles of R-CHOP21 / 2-3 cycles of R-HAD28 (alternating)
* Patients with serious underlying medical conditions, which could impair the ability to receive maintenance treatment
* Calculated creatinine clearance of < 30 mL / min
* ANC is < 1,000 cells/mm³
* Platelet count is < 50,000 cells/mm³

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2.5 years
  2.5 years after last patient randomized in maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dreyling, Prof. Dr., Principal Investigator — MCL Network; Vincent Ribrag, Dr, Principal Investigator — Lymphoma Study Association; Johanna Cornelia Kluin-Nelemans, Prof. Dr., Principal Investigator — MCL Network
Locations (143):
- Belgium (9):
  - ZNA Stuivenberg, Antwerp
  - A. Z. Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Université Catholique de Louvain Saint Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - AZ Groeninge, Kortrijk
  - CHU de Liège, Liège
  - CH de la Tourelle-Peltzer, Verviers
  - Université Catholique de Louvain Mont Godinne, Yvoir
- France (56):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH d Avignon - Hopital Henri Duffaut, Avignon
  - CH Côte Basque, Bayonne
  - CHU Jean Minjoz, Besançon
  - CH de Blois, Blois
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - CH du Dr Duchenne, Boulogne-sur-Mer
  - CHU Morvan, Brest
  - CHU Caen, Caen
  - MEDIPOLE de SAVOIE, Challes-les-Eaux
  - CH Chambéry, Chambéry
  - CHU de Châlon-sur-Sâone - William Morey, Châlon-sur-Sâone
  - Hopital Antoine Beclere, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Pôle Santé République, Clermont-Ferrand
  - CH Sud Francilien de Corbeil, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - CHU Le Bocage, Dijon
  - CH Dunkerque, Dunkirk
  - Institut Daniel Hollard, Grenoble
  - CHU de Grenoble, Grenoble
  - CH Départemental, La Roche-sur-Yon
  - Groupe Hospitalier La Rochelle - Ré - Aunis, La Rochelle
  - Hôpital André Mignot, Le Chesnay
  - CH du Mans, Le Mans
  - Clinique Victor Hugo, Le Mans
  - CH de Lens, Lens
  - CHU Claude Hurriez, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - CH de Meaux, Meaux
  - Hôpital Bon Secours, Metz
  - CH de la Région Annecy-Genevois, Metz-Tessy
  - CHU Montpellier, Montpellier
  - CHU Hôtel Dieu, Nantes
  - CHR de la Source, Orléans
  - Hopital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Necker, Paris
  - CH Perpignan, Perpignan
  - Hôpital Haut Lévêque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CH de Quimper Cornouaille, Quimper
  - CHU Robert Debre, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de cancérologie de la Loire, Saint-Priest-en-Jarez
  - CH Saint Quentin, Saint-Quentin
  - CHU de Strasbourg, Strasbourg
  - CHU Purpan, Toulouse
  - CHU Bretonneau, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (35):
  - Gesundheitszentrum St. Marien GmbH, Amberg
  - Charite´ Universitätsmedizin Berlin Campus Benjamin Franklin, Berlin
  - Charite´Universitätsmedizin Berlin Campus Virchow-Klinikum, Berlin
  - Städt. Klinikum Braunschweig gGmbH, Braunschweig
  - DIAKO Ev. Diakonie-Krankenhaus gemeinnützige GmbH, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Marien Hospital Düsseldorf, Düsseldorf
  - St. Antonius Hospital, Eschweiler
  - Universitätsklinikum Essen, Essen
  - Klinikum Frankfurt GmbH, Frankfurt (Oder)
  - Universitätsmedizin Greifswald, Greifswald
  - Kath. Krankenhaus Hagen gem. GmbH, Hagen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum Herford, Herford
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Städt. Klinikum Karlsruhe, Karlsruhe
  - Uni-Klinikum-Schleswig-Holstein im Städt. Krankenhaus Kiel, Kiel
  - Internistische Praxis /Hämatologie und Onkologie, Kronach
  - Onkologisches Zentrum - Lebach, Lebach
  - Klinikum Ludwigshafen, Ludwigshafen
  - Kliniken Maria Hilf GmbH (Krankenhaus St. Franziskus), Mönchengladbach
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Klinikum rechts der Isar der TU München, München
  - Klinikum der Universität München, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Universitätsklinikum Münster, Münster
  - Gemeinschaftspraxis für Hämatologie und internistische Onkologie, Neumarkt
  - Klinikum Nürnberg, Nuremberg
  - Gemeinschaftspraxis für Innere Medizin, Hämatologie und internistische Onkologie, Offenbach
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Universitätsklinik Rostock, Rostock
  - Mutterhaus der Borromäerinnen GmbH, Trier
  - University Hospital Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Netherlands (25):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - MC Alkmaar, Alkmaar
  - VUMC, Amsterdam
  - OLVG, Amsterdam
  - AMC, Amsterdam
  - Amphia ziekenhuis, locatie Langendijk, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Gemini Ziekenhuis, Den Helder
  - Medisch Spectrum Twente, Enschede
  - Zuyderland MC, Geleen
  - Admiraal De Ruyter Ziekenhuis, Goes, Goes
  - Groene Hart Ziekenhuis, Gouda
  - UMCG, Groningen
  - Spaarne ziekenhuis, Hoofddorp
  - MC Leeuwarden Zuid, Leeuwarden
  - Maastricht UMC, Maastricht
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Radboudumc, Nijmegen
  - Bravis ziekenhuis, Roosendaal
  - Erasmus MC - Centrum, Rotterdam
  - Erasmus MC - Daniel, Rotterdam
  - Maasstadziekenhuis, Rotterdam
  - Hagaziekenhuis, locatie Leyweg, The Hague
  - St.Elisabeth ZH, Tilburg
  - Isala Klinieken, Sophia, Zwolle
- Poland (6):
  - Gdansk University School of Medicine, Gdansk
  - Szpitale Wojewódzkie, Gdynia
  - University Hospital, Krakow
  - Warminsko-Mazurskie Centrum Onkologii, Olsztyn
  - Institute of Hematology and Transfusiology, Warsaw
  - MSCM Institute and Oncology Centre, Warsaw
- Instituto Português de Oncologia de Lisboa de Francisco Gentil, Lisbon, Portugal
- Spain (11):
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Institut Catala d'Oncologia (ICO) - Hospital Germans Trias y Pujol, Badalona
  - Hospital Universitario Vall d'hebron, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Clinico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No